CLINICAL TRIAL: NCT00278382
Title: A Phase 2 Study of BAY 43-9006 (IND 69896) in Chemosensitive Relapsed Aggressive Non-Hodgkin's Lymphomas
Brief Title: Sorafenib in Treating Patients With Recurrent Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02682; GCC0508; CDR0000456442 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Anaplastic Large Cell Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell | interventions — Sorafenib

ARMS (1):
- Treatment (sorafenib tosylate) (Experimental): Patients receive oral sorafenib twice daily in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sorafenib tosylate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: sorafenib tosylate — Given orally
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Sorafenib may stop the growth of cancer cells by blocking blood flow to the cancer and by blocking some of the enzymes needed for cell growth. This phase II trial is studying how well sorafenib works in treating patients with chemosensitive recurrent aggressive non-Hodgkin's lymphoma

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the overall response rate, including complete and partial responses, in patients with chemosensitive, relapsed, aggressive, non-Hodgkin's lymphoma treated with sorafenib.

SECONDARY OBJECTIVES:

I. Determine progression-free and overall survival of patients treated with this drug.

II. Determine response duration in patients treated with this drug.

OUTLINE: This is an open-label study.

Patients receive oral sorafenib twice daily in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 33 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed aggressive* non-Hodgkin's lymphoma by excisional-node biopsy or core needle biopsy and bone marrow biopsy, including 1 of the following types:

  * Mantle cell lymphoma
  * Primary mediastinal large B-cell lymphoma
  * Diffuse large B-cell lymphoma
  * Anaplastic large cell lymphoma (T-cell or null-cell type)
* Recurrent disease
* Patients must have received ≥ 1 induction regimen containing anthracyclines (e.g., CHOP [with or without rituximab] or R-EPOCH)
* Chemosensitive disease at the time of relapse

  * Patients who responded with a complete or partial remission that lasted at least 8 weeks after their last chemotherapy regimen are considered chemosensitive
* Measurable disease, defined as a lymph node or a nodal mass of > 1 cm in its longest transverse diameter on CT scan
* Ineligible for, refused, or relapsed after stem cell transplant (for patients with non-mantle cell lymphoma)
* No known brain metastases, including meningeal involvement
* ECOG performance status (PS) 0-2
* Karnofsky PS 60-100%
* Life expectancy > 3 months
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* Fertile patients must use effective contraception
* Not pregnant or nursing
* Negative pregnancy test
* No uncontrolled illness
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to sorafenib
* No known positive HIV serology
* No inflammatory bowel disease
* No swallowing dysfunction that would prevent ingestion of pills
* No hemorrhagic diathesis
* No ongoing or active infection
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No uncontrolled hypertension
* No psychiatric or social situation that would limit compliance with study requirements
* No poorly controlled medical condition that would seriously complicate compliance with this study
* Patients with inflammatory or exfoliative skin disease are excluded (regardless of the extent of the involvement) unless the skin condition is lymphoma related
* See Disease Characteristics
* Previous treatment-related toxic effects should be resolved to grade 1 or better
* No chemotherapy or radiation therapy within the past 4 weeks

  * 6 weeks for nitrosoureas or mitomycin C
* No prior antibody therapy for at least 3 months
* Prior radiation for localized disease or total body irradiation as part of a conditioning regimen prior to stem cell transplant allowed
* Prior radio-immunotherapy allowed
* No concurrent therapeutic anticoagulation

  * Prophylactic anticoagulation (i.e., low-dose warfarin) of venous or arterial access devices are acceptable provided that the requirements for PT, INR, and PTT are met
* No concurrent use of another investigational agent
* No concurrent use of the following drugs: phenytoin, carbamazepine, phenobarbital, rifampin, or Hypericum perforatum (St. John's wort)
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2005-10; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Objective response rate (complete and partial response) | Up to 2 years
  Will be calculated as the percent of evaluable patients whose best response is a CR or PR. The exact binomial method will be used to determine the confidence interval of response rate.

SECONDARY OUTCOMES:
Overall survival | Up to 2 years
  The Kaplan-Meier product-limit method will be used in analysis of survival time.
Time to disease progression | Up to 2 years
  The Kaplan-Meier product-limit method will be used in analysis of time to disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Meyer Heyman, Principal Investigator — University of Maryland Greenebaum Cancer Center
Locations (1):
- University of Maryland Greenebaum Cancer Center, Baltimore, Maryland, United States